CLINICAL TRIAL: NCT06441773
Title: Impact of Respiratory Rehabilitation on Quality of Life in Patients With Metastatic Non-small Cell Lung Cancer Treated With Immunotherapy and Chemotherapy in the Maintenance Phase
Acronym: REHABIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC22.0255; 2024-A02083-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: Respiratory rehabilitation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A two-center, randomized, open-label, parallel-group, ratio-distributed (1:1) trial comparing the impact of respiratory rehabilitation (RR) on quality of life at 2 months in patients with advanced NSCLC associated with RR versus patients with advanced NSCLC without RR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Maintenance of chemotherapy and immunotherapy alone: without respiratory rehabilitation (control group)
- Respiratory rehabilition (Experimental): Maintenance of chemotherapy and immunotherapy combined with a respiratory rehabilitation program of 2 sessions per week for 8 weeks (respiratory rehabilitation group) = 16 sessions
  Interventions: Procedure: Respiratory Rehabilitation

INTERVENTIONS:
Procedure: Respiratory Rehabilitation — An initial assessment is conducted upon admission to personalize the program. This includes:
  Clinical examination Spirometry Maximum Inspiratory Pressure (PImax) measurement Multidimensional Dyspnea Profile questionnaire at end of TM6 Exercise Functional Testing Measurement of quadriceps strength and endurance Blood gases Educational interview and shared educational assessment London Chest Activity of Daily Living (LCADL) Tobacco and/or dietary consultation
  The respiratory rehabilitation program, performed twice a week, includes:
  Exercise training on an ergocycle and treadmill (30 minutes at ventilatory threshold for the ergocycle; 30 minutes at 60-80% walking speed for the treadmill; or dyspnea rated 4-6 on the Borg scale after endurance exercise) Quadriceps muscle strengthening Therapeutic education program Group gymnastics Smoking cessation assistance Socio-psychological and nutritional support
  Arms: Respiratory rehabilition

SUMMARY:
Lung cancer is highly prevalent, with approximately 46,363 new cases in 2018, accounting for 20.6% of cancer deaths in France. At diagnosis, 70% of patients have advanced or metastatic cancer, treatable only by palliative care. Respiratory rehabilitation aims to reduce symptoms, enhance performance, increase autonomy, and improve patients' quality of life. While effective for COPD patients and other conditions causing dyspnea, its benefits in advanced, non-operable lung cancer are less studied. Some studies have shown the feasibility and safety of respiratory rehabilitation, but few have compared its impact on non-operable lung cancer patients or assessed its effect on quality of life. The main objective of the proposed study is to evaluate the impact of a respiratory rehabilitation program on the quality of life of patients with non-small cell lung cancer (NSCLC) undergoing maintenance chemotherapy and immunotherapy, compared to a control group receiving standard care.

DETAILED DESCRIPTION:
Lung cancer accounts for an estimated 46,363 new cases in 2018. At the time of diagnosis, 70% of patients have locally advanced or metastatic cancer that can no longer be treated by surgery, but only by palliative therapy. It is the 4th most common cancer in France, and the most common worldwide. Lung cancer accounts for 20.6% of all cancer deaths in France.

Respiratory rehabilitation aims to minimize symptoms linked to the underlying pathology, and to enhance performance, increase autonomy and promote activities of daily living. It also aims to improve health-related quality of life and long-term maintenance of behavioral changes. It has been shown to be effective for COPD patients. Respiratory rehabilitation has also demonstrated its benefits in other pathologies whose common denominator is dyspnea, such as interstitial lung disease and pulmonary hypertension. In the case of operable lung cancers, numerous studies have focused on the preoperative and postoperative benefits.

Very few studies have focused on its benefits in advanced, non-operable lung cancer.

The team of Olivier et al. studied the benefits of home respiratory rehabilitation for 8 weeks in patients with advanced or metastatic lung cancer or mesothelioma treated with concomitant chemotherapy. Their study shows feasibility and safety for patients who complete the program, but the authors point out that the absence of a control arm and the small number of patients mean that the benefits of respiratory rehabilitation cannot be confirmed.

The team of Edbrooke et al., in 2019, is studying the value of a home-based rehabilitation program. The aim of the study is to demonstrate the efficacy of respiratory rehabilitation compared with standard care, a randomized controlled superiority trial. The study showed no statistically significant difference at 9 weeks on the primary endpoint (the 6-min walk test), due to a lack of power in the trial. A final study (Park et al.) showed the feasibility of outpatient rehabilitation in twelve patients, but did not conclude on the value of respiratory rehabilitation.

Thus, while a few studies have demonstrated the feasibility of respiratory rehabilitation in patients with bronchial cancer, few comparative studies have evaluated the impact of rehabilitation in patients with non-operable bronchial cancer, and no study has assessed the impact of respiratory rehabilitation on quality of life (as a primary endpoint), although this would appear to be an essential element in the care of these patients.

The main objective of our study is to evaluate the impact of a respiratory rehabilitation program (rehabilitation group) in patients with non-small cell lung cancer (NSCLC) treated with chemotherapy and immunotherapy in the maintenance phase compared with patients with NSCLC treated with chemotherapy and immunotherapy in the maintenance phase (control group), on quality of life at 2 months (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage IV non-small cell lung cancer patient
* First-line treatment with chemotherapy combined with immunotherapy in the maintenance phase
* Adenocarcinoma patient: maintenance with Alimta combined with pembrolizumab
* Squamous cell carcinoma patient: maintenance with pembrolizumab alone
* Age of at least 18 years
* Performance status of 0 or 1
* Estimated life expectancy > 12 weeks
* No contraindications to respiratory rehabilitation
* Adequate organ function, demonstrated by laboratory results within the last 3 weeks, allowing maintenance treatment:
* Normal liver function: bilirubin < 1.5 x ULN, ALT and AST < 2.5 x ULN or < 5 x ULN in the case of liver metastases.
* Renal function (creatinine clearance calculation of at least > 45 mL/min).
* Hematological function: absolute neutrophil count > 1.5 x 10^9/L and/or platelets > 100 x 10^9/L, hemoglobin > 8 g/dL.
* Informed consent to participate in the study must be signed
* Patient must be affiliated with or beneficiary of social security

Exclusion Criteria:

* Small cell lung cancer, mesothelioma, neuroendocrine lung cancer
* Patients with orthopedic disorders preventing respiratory rehabilitation that, in the investigator's opinion, could interfere with respiratory rehabilitation
* Unresolved toxicity from previous treatment of grade > 1 (except alopecia) that, in the investigator's opinion, could interfere with respiratory rehabilitation
* Symptomatic brain metastases (corticosteroid treatment is allowed if the doses administered are stable for at least one month before inclusion)
* Bone metastases preventing respiratory rehabilitation
* Contraindication to respiratory rehabilitation
* Uncontrolled infection
* Pregnancy and breastfeeding
* Surgery within two months prior to inclusion that could interfere with respiratory rehabilitation
* Persons under legal protection (guardianship or curatorship) or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Measurement Using EORTC QLQ-C30 | Week 0
  The primary endpoint is the measurement of quality of life, assessed by the composite score from the sum of EORTC QLQ-C30. The evaluation will be conducted by filling out the quality of life questionnaires at inclusion (=Week 0) and at 8 weeks
Quality of Life Measurement Using EORTC QLQ-LC13 | Week 0
  The primary endpoint is the measurement of quality of life, assessed by the composite score from the sum of EORTC QLQ-LC13. The evaluation will be conducted by filling out the quality of life questionnaires at inclusion (=Week 0) and at 8 weeks
Quality of Life Measurement Using EORTC QLQ-C30 | Week 8
  The primary endpoint is the measurement of quality of life, assessed by the composite score from the sum of EORTC QLQ-C30. The evaluation will be conducted by filling out the quality of life questionnaires at inclusion (=Week 0) and at 8 weeks
Quality of Life Measurement Using EORTC QLQ-LC13 | Week 8
  The primary endpoint is the measurement of quality of life, assessed by the composite score from the sum of EORTC QLQ-LC13. The evaluation will be conducted by filling out the quality of life questionnaires at inclusion (=Week 0) and at 8 weeks

SECONDARY OUTCOMES:
Evaluation of quality of life using multiple modalities of the QLQ-C30. | Week 0
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C30 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C30. | Week 8
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C30 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C30. | Month 6
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C30 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C30. | Month 12
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C30 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C13. | Week 0
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C13 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C13 | Week 8
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C13 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C13 | Month 6
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C13 questionnaire.
Evaluation of quality of life using multiple modalities of the QLQ-C13 | Month 12
  Quality of life measurement using the functional scales and symptom scales of the QLQ-C13 questionnaire.
Evaluation of quality of life using the global health score of the QLQ-C30 | Month 6
  Quality of life measurement using the global health score of the QLQ-C30 at 6 months and 1 year.
Evaluation of quality of life using the global health score of the QLQ-C30 | Month 12
  Quality of life measurement using the global health score of the QLQ-C30 at 6 months and 1 year.
Evaluation of the number of deceased and surviving patients throughout the study follow-up. | Week 8
  Evaluation of the number of deceased and surviving patients throughout the study follow-up.
Evaluation of the number of deceased and surviving patients throughout the study follow-up. | Month 6
  Evaluation of the number of deceased and surviving patients throughout the study follow-up.
Evaluation of the number of deceased and surviving patients throughout the study follow-up. | Month 12
  Evaluation of the number of deceased and surviving patients throughout the study follow-up.
Study of tumor response evaluation | Week 8
  Measurement of median Progression-Free Survival (based on RECIST criteria = tumor response evaluation) throughout the study follow-up.
Study of tumor response evaluation | Month 6
  Measurement of median Progression-Free Survival (based on RECIST criteria = tumor response evaluation) throughout the study follow-up.
Study of tumor response evaluation | Month 12
  Measurement of median Progression-Free Survival (based on RECIST criteria = tumor response evaluation) throughout the study follow-up.
Evaluation of exercise capacity using 6-Minute Walk Test | Week 0
  Measurement of exercise capacity using the 6-Minute Walk Test (6MWT) at Week 0 and at 8 weeks (after 16 sessions for the respiratory rehabilitation group)
Evaluation of exercise capacity using 6-Minute Walk Test | Week 8
  Measurement of exercise capacity using the 6-Minute Walk Test (6MWT) at Week 0 and at 8 weeks (after 16 sessions for the respiratory rehabilitation group)
Evaluation of the number of events of interest | Week 8
  Evaluation of the number of events of interest
Evaluation of the number of events of interest | Month 6
  Evaluation of the number of events of interest
Evaluation of the number of events of interest | Month 12
  Evaluation of the number of events of interest
Evaluation of the number of hospitalizations | Week 8
  Number of hospitalizations other than for maintenance treatment
Evaluation of the number of hospitalizations | Month 6
  Number of hospitalizations other than for maintenance treatment
Evaluation of the number of hospitalizations | Month 12
  Number of hospitalizations other than for maintenance treatment
Evaluation of anxiety and depressive disorders | Week 0
  Measurement of anxiety and depressive disorders (HAD questionnaire) between Week 0 and Week 8
Evaluation of anxiety and depressive disorders | Week 8
  Measurement of anxiety and depressive disorders (HAD questionnaire) between Week 0 and Week 8
Evaluation of dyspnea with mMRC scale | Week 0
  Evaluation of dyspnea (MMRC scale) at Week 0 and at 8 weeks
Evaluation of dyspnea with mMRC scale | Week 8
  Evaluation of dyspnea (MMRC scale) at Week 0 and at 8 weeks
Evaluation of dyspnea with Dyspnea-12 questionnaire | Week 0
  Evaluation of dyspnea (Dyspnea-12 questionnaire) at Week 0 and at 8 weeks
Evaluation of dyspnea with Dyspnea-12 questionnaire | Week 8
  Evaluation of dyspnea (Dyspnea-12 questionnaire) at Week 0 and at 8 weeks
Evaluation of self-esteem with ISP-6 questionnaire | Week 0
  Evaluation of self-esteem (ISP-6 questionnaire) at Week 0 and at 8 weeks
Evaluation of self-esteem with ISP-6 questionnaire | Week 8
  Evaluation of self-esteem (ISP-6 questionnaire) at Week 0 and at 8 weeks
Evaluation of tiredness with EORTC QLQ FA-12 questionnaire | Week 8
  Evaluation of tiredness (EORTC QLQ FA-12 questionnaire) at Week 0 and at 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Brest, Brest
  - CH Morlaix, Morlaix
  - CH Cornouaille, Quimper